CLINICAL TRIAL: NCT02014207
Title: The Effect of Potato Fries Processing on Food Intake, Satiety and Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Purpose: Prevention
Other Study IDs: Potato study 1: processing; OMAFRA (Other Grant/Funding Number: SR9174)
Record Dates: First submitted 2013-12-07; First posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Obesity; Overweight; Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus; Metabolic Syndrome

ARMS (5):
- golden crinkle (Experimental)
  Interventions: Other: dietary treatment
- high blanch (Experimental)
  Interventions: Other: dietary treatment
- low blanche (Experimental)
  Interventions: Other: dietary treatment
- high chill (Experimental)
  Interventions: Other: dietary treatment
- low chill (Experimental)
  Interventions: Other: dietary treatment

INTERVENTIONS:
Other: dietary treatment

SUMMARY:
Potato is one of the world's most popular foods and is widely accepted as a staple food. The objective of this study is to determine the effect of altering commercial blanching and cooling times during manufacture of frozen fries produced by the on blood glucose, satiety and appetite. It hypothesized that the processing regime predetermines the physiologic responses to ingested product and therefore it is possible to produce healthier product lines of potato fries.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men with a body mass index (kg/m2) of 20-24.9

Exclusion Criteria:

* smocking, medication, breakfast skipping, restrained eating

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Dates: Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
blood glucose | 120 min
  Glycaemic response will be measured before the treatment (baseline) and at 15, 30, 45, 60, 90 and 120 min after the treatment. The glucose concentration will be measured in capillary blood using portable glucose meter.

SECONDARY OUTCOMES:
food intake | 120 min
  Ad libidum food intake will be measure at 120 min using test pizza meal. The amount of consumed test meal (g) will be converted to the energy (kcal).

OTHER OUTCOMES:
subjective appetite | 120 min
  Subjective appetite will be measured with visual analogue scales at 0 min immediately before the treatment (baseline) and at 15, 30, 45, 60, 90 and 120 min after the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutritional Sciences, Toronto, Ontario, Canada